CLINICAL TRIAL: NCT01642953
Title: Prospective Clinical Study for Early Recovery After Gastric Cancer Surgery
Brief Title: Early Recovery After Gastric Cancer Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Collaborators: JW Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Hoon Hur, Assistant Professor, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-MED-MDB-12-002
Record Dates: First submitted 2012-07-14; First posted 2012-07-17 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Fasting; Malignant Neoplasm of Stomach
Keywords: Gastric cancer surgery; Early oral feeding; Fast track surgery
MeSH Terms: conditions — Fasting; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Early recovery (Experimental): Patients who enroll in this arm are supplied a liquid diet one day before surgery without bowel preparation.
  After gastric cancer surgery, they start sips of water on postoperative first day, and they are discharged once they exhibit at least three times soft diet without specific complaint and had normal clinical status and physical examination.
  Interventions: Dietary Supplement: Early recovery

INTERVENTIONS:
Dietary Supplement: Early recovery — The patients are started on sips of water on the first postoperative day. If they are tolerable, a liquid diet is started on the second postoperative day, and a soft diet on a third postoperative day for them. We have a plan to discharge the patients on the fourth postoperative day if they exhibit at least three times soft diet without specific complaint and had normal clinical status and physical examination.

SUMMARY:
Study preparation

* To progress this prospective study, the investigators analyzed the retrospective data of 426 patients who had been managed with conventional critical pathway after gastric cancer surgery during last 1 year.
* Through this retrospective analysis, we decided the inclusion criteria which showed significantly the lower complication rate and shorter hospital stay.

Method for Prospective study

* Patients who enroll in this prospective study are administered and are supplied a liquid diet one day before surgery without bowel preparation.
* After gastric cancer surgery, they start sips of water on postoperative first day, and they are discharged once they exhibit at least three times soft diet without specific complaint and had normal clinical status and physical examination.

DETAILED DESCRIPTION:
Enrollment of patients

* Before the patients are enrolled in this study, they give us informed consents.
* A liquid diet is supplied beginning from the morning of the day prior to operation to the midnight.

Operation and postoperative management

* All procedures are approached by laparoscopic surgery, and partial gastrectomy with lymph node dissection are performed.
* The patients who are considered to be difficult to progress early oral feeding in surgical field are excluded from the study.
* Nasogastric tube is not applied to patients.
* Postoperative pain is managed by non-opioid pain killer.
* The patients are started on sips of water on the first postoperative day.
* If they are tolerable, a liquid diet is started on the second postoperative day, and a soft diet on a third postoperative day for them.
* We have a plan to discharge the patients on the fourth postoperative day if they exhibit at least three times soft diet without specific complaint and had normal clinical status and physical examination.

Evaluation of patients

- The patients are followed up to 30 days after discharge from hospital, and we check whether they are tolerable without any compliant and are readmitted.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with gastric adenocarcinoma
* 65 years old and blew
* Patients are expected to be undergone distal subtotal gastrectomy
* No complication by gastric cancer
* No synchronous metastatic lesions
* Laparoscopic or robotic surgery
* Informed consent

Exclusion Criteria:

* Previous gastrectomy history
* Combined surgery due to synchronous malignancy
* Patients with major organ dysfunction

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Drop rate from critical pathway | 4 days
  It is defined as the proportion of dropped patients from 4 days critical pathway

SECONDARY OUTCOMES:
Postoperative pain | 7 days
  It is defined as the change of pain scale after surgery
Postoperative complication | 30 days
  It is defined the complications after surgery
Postoperative mortality | 30 days
  It will defined as the death case during 30 days after surgery
Recovery after surgery | 7 days
  It is defined as the time to first flatus and recovery of bowel activity after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hoon Hur, Prof., Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, South Korea

REFERENCES:
- [Derived] Roh CK, Son SY, Lee SY, Hur H, Han SU. Clinical pathway for enhanced recovery after surgery for gastric cancer: A prospective single-center phase II clinical trial for safety and efficacy. J Surg Oncol. 2020 Mar;121(4):662-669. doi: 10.1002/jso.25837. Epub 2020 Jan 12. PMID 31930513